CLINICAL TRIAL: NCT06184113
Title: Comparison of Apixaban and Aspirin for the Prevention of Latent Bioprosthetic Valve Thrombosis After Aortic Valve Replacement Surgery: Study Protocol for a Prospective Randomized Trial
Brief Title: Apixaban for the Prevention of Latent Biological Valve Thrombosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Tomislav Kopjar, Principal Investigator, Clinical Hospital Centre Zagreb
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8.1-23/77-3; 02/013 AG
Record Dates: First submitted 2023-12-03; First posted 2023-12-28 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Aortic Valve Replacement; Antithrombotic Therapy; Bioprosthetic Valve Thrombosis; Rapid Deployment Valves
MeSH Terms: interventions — Tomography, X-Ray Computed; Echocardiography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Patients randomised to the intervention arm will receive an open-label dose adjusted apixaban twice a day. The treatment will be continued for three months. After the tree-month treatment period apixaban will be stopped and acetylsalicylic acid will be started.
  Interventions: Procedure: Aortic valve replacement surgery; Diagnostic Test: Computed tomography; Diagnostic Test: Echocardiography
- Control Arm (Active Comparator): Patients assigned to the control arm will receive an open-label low dose acetylsalicylic acid indefinitely.
  Interventions: Procedure: Aortic valve replacement surgery; Diagnostic Test: Computed tomography; Diagnostic Test: Echocardiography

INTERVENTIONS:
Procedure: Aortic valve replacement surgery — Patients undergoing first-time isolated aortic valve replacement with a rapid deployment biological prosthesis.
Diagnostic Test: Computed tomography — All the study patients will undergo a computed tomography imaging to assess for hypo-attenuated leaflet thickening and reduced leaflet mobility of the biological prosthesis following the three-month treatment period.
Diagnostic Test: Echocardiography — All the study patients will undergo a transthoracic echocardiography before hospital discharge and following the three-month treatment period.

SUMMARY:
Background: The optimal antithrombotic strategy early after aortic valve replacement surgery with a biological valve remains controversial due to lack of high-quality evidence. Either oral anticoagulants or acetylsalicylic acid should be considered for the first three months. Hypo-attenuated leaflet thickening on cardiac compute tomography has been associated with latent bioprosthetic valve thrombosis and may be prevented with anticoagulation. The investigators hypothesize that anticoagulation with apixaban is superior to single antiplatelet therapy with acetylsalicylic acid in reduction of hypo-attenuated leaflet thickening of bioprosthetic valves after aortic valve replacement.

Methods: In this prospective, open-label, randomized trial patients without an indication for oral anticoagulation undergoing isolated aortic valve replacement surgery with novel rapid-deployment bioprosthetic valves will be randomized. The treatment group will receive 5 mg of apixaban twice a day for the first three months and 100 mg of acetylsalicylic acid thereafter. The control group will have 100 mg of acetylsalicylic acid once a day indefinitely. After the three-month treatment period a contrast enhanced electrocardiogram-gated cardiac computed tomography will be performed to identify hypo-attenuated leaflet thickening of the bioprosthetic valve. The primary objective of the study is to assess possible superiority of the treatment group in the prevention of hypo-attenuated leaflet thickening three months after randomization. Secondary objective is to assess possible noninferiority for safety of apixaban-based strategy when compared to acetylsalicylic acid at three months.

Discussion: Antithrombotic therapy after aortic valve replacement surgery is used to prevent valve thrombosis and systemic thromboembolism. Latent bioprosthetic valve thrombosis is a precursor of clinically significant prosthetic valve dysfunction or thromboembolic event. The hallmark feature of latent bioprosthetic valve thrombosis is hypo-attenuated leaflet thickening on cardiac computed tomography. Subclinical leaflet thrombosis occurs frequently in bioprosthetic aortic valves, more commonly in transcatheter than in surgical valves. There is no evidence on the effect of direct oral anticoagulants on the incidence of hypo-attenuated leaflet thickening after surgical aortic valve replacement with rapid deployment bioprostheses.

ELIGIBILITY:
Inclusion Criteria

* Men and women aged 65 or older with aortic valve stenosis undergoing successful isolated first-time aortic valve replacement with a rapid deployment bioprosthetic valve
* Signed informed consent to participate in the research

Exclusion Criteria:

* Indication for long-term use of anticoagulant therapy
* Indication for dual antiplatelet therapy
* Contraindication to anticoagulation or antiplatelet therapy
* Inability to start the study drug within the planned randomization period
* History of atrial fibrillation
* Known hemorrhagic diathesis
* Presence of other significant heart pathology
* Prior open-heart surgery
* Presence of liver failure or other coagulopathy
* Aortic valve infective endocarditis
* Severe renal failure
* Allergy to iodine contrast

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with hypo-attenuated leaflet thickening | At the end of treatment at 3 months
  Hypo-attenuated leaflet thickening is identified as increased thickness of one or more leaﬂets of the bioprosthetic valve on contrast-enhanced electrocardiogram gated cardiac computed tomography. Grade 3 on a 4-tier semiquantitative grading scale describes more than 50% and less than 75% of leaflet involvement. Grade 3 or higher of hypo-attenuated leaflet thickening of at least one bioprosthetic valve leaflet will be considered.

SECONDARY OUTCOMES:
Proportion of patients with bleeding, thromboembolic event, or death | From enrolment to the end of treatment at 3 months
  The safety composite outcome will be comprised of all types of VARC-3 bleeding events, thromboembolic events (myocardial infarction and stroke), and death from any cause.

OTHER OUTCOMES:
Rate of hypo-attenuated leaflet thickening | At the end of treatment at 3 months
  Hypo-attenuated leaflet thickening is identified as increased thickness of one or more leaﬂets of the bioprosthetic valve on contrast-enhanced electrocardiogram gated cardiac computed tomography. Grade 3 on a 4-tier semiquantitative grading scale describes more than 50% and less than 75% of leaflet involvement which will be considered significant. Grade 3 or higher will be considered significant.
Rate of reduced leaflet mobility | At the end of treatment at 3 months
  Leaflet restriction caused by hypo-attenuated leaflet thickening can be described as reduced leaflet mobility. Using computed tomography, reduced leaflet motion will be assessed on short-axis reformatted images during systole and 4D volume rendering images. The extent can be described per leaﬂet, using a 4-tier grading scale in systole: (1) not present, (2) < 50% restriction in leaflet excursion, (3) ≥50% restriction in leaflet excursion and (4) immobile leaflet. Grade 3 or higher will be considered significant.
Proportion of patients in each NYHA functional class | At the end of treatment at 3 months
  New York Heart Association functional classification of heart failure. Class I, no limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation or shortness of breath. Class II, slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain. Class III, marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain. Class IV, symptoms of heart failure at rest. Any physical activity causes further discomfort.
Rates of bioprosthetic valve deterioration | At the end of treatment at 3 months
  Stage 1 is described with morphological valve deterioration without significant hemodynamic changes. Stage 2 is characterized with moderate hemodynamic valve deterioration with an increase in mean transvalvular gradient ≥10 mmHg, and Stage 3 with severe hemodynamic valve deterioration with an increase in mean transvalvular gradient ≥20 mmHg.
Rate of VARC-3 bleeding events | From enrolment to the end of treatment at 3 months
  A descriptive classification scheme for VARC-3 bleeding, like the Bleeding Academic Research Consortium classification has been proposed. It includes 4-type bleeding scale: Type 1 (minor), Type 2 (major), Type 3 (life-threatening), and Type 4 (leading to death) bleeding.
Proportion of patients with myocardial infarction | From enrolment to the end of treatment at 3 months
  Myocardial infarction with elevated biomarkers cTn values with at least symptoms of acute ischaemia, new ischaemic ECG changes, new pathologic Q-waves, imaging evidence of a new loss of viable myocardium or new wall motion abnormality, identification of a coronary thrombus by angiography or autopsy.
Proportion of patients with stroke | From enrolment to the end of treatment at 3 months
  All stroke (ischaemic stroke, haemorrhagic stroke, or any stroke not otherwise specified) with signs and symptoms and with pathology or neuroimaging evidence of central nervous system infarction, or absence of other apparent causes.
Proportion of patients that died | From enrolment to the end of treatment at 3 months
  All cause mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Tomislav Kopjar, MD, PhD, Principal Investigator — Clinical Hospital Centre Zagreb
Locations (1):
- University Hospital Center Zagreb, Zagreb, Croatia

REFERENCES:
- [Derived] Kopjar T, Gasparovic H, Paar MH, Lovric D, Cerina P, Tokic T, Milicic D. Comparison of apixaban versus aspirin for the prevention of latent bioprosthetic aortic valve thrombosis: study protocol for a prospective randomized trial. Trials. 2024 May 16;25(1):324. doi: 10.1186/s13063-024-08175-w. PMID 38755709